CLINICAL TRIAL: NCT01816113
Title: A Phase Ia Clinical Trial to Assess the Safety and Immunogenicity of New Plasmodium Vivax Malaria Vaccine Candidates ChAd63 PvDBP Alone and With MVA PvDBP
Brief Title: Phase Ia Study of ChAd63/MVA PvDBP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC051
Record Dates: First submitted 2013-03-13; First posted 2013-03-21 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Malaria; Plasmodium Vivax
Keywords: PvDBP; Malaria; Plasmodium vivax
MeSH Terms: conditions — Malaria; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 4 volunteers; 1 dose of ChAd63 PvDBP 5 x 10^9 vp intramuscularly
  Interventions: Biological: ChAd63 PvDBP 5 x 10^9
- Group 2A (Experimental): 4 volunteers; 1 dose of ChAd63 PvDBP 5 x 10^10 vp intramuscularly
  Interventions: Biological: ChAd63 PvDBP 5 x 10^10
- Group 2B (Experimental): 8 volunteers; 1 dose of ChAd63 PvDBP 5 x 10^10 vp intramuscularly and 1 dose MVA PvDBP 1 x 10^8 pfu 8 weeks later intramuscularly
  Interventions: Biological: ChAd63 PvDBP 5 x 10^10; Biological: MVA PvDBP 1 x 10^8
- Group 2C (Experimental): 8 volunteers; 1 dose of ChAd63 PvDBP 5 x 10^10 vp intramuscularly and 1 dose MVA PvDBP 2 x 10^8 pfu 8 weeks later intramuscularly
  Interventions: Biological: ChAd63 PvDBP 5 x 10^10; Biological: MVA PvDBP 2 x 10^8

INTERVENTIONS:
Biological: ChAd63 PvDBP 5 x 10^9 — 1 dose of ChAd63 PvDBP 5 x 10^9 vp intramuscularly
  Arms: Group 1
Biological: ChAd63 PvDBP 5 x 10^10 — 1 dose of ChAd63 PvDBP 5 x 10^10 vp intramuscularly
  Arms: Group 2A; Group 2B; Group 2C
Biological: MVA PvDBP 1 x 10^8 — 1 dose MVA PvDBP 1 x 108 pfu 8 weeks later intramuscularly
  Arms: Group 2B
Biological: MVA PvDBP 2 x 10^8 — 1 dose MVA PvDBP 2 x 108 pfu 8 weeks later intramuscularly
  Arms: Group 2C

SUMMARY:
This is an open label phase Ia study, to assess the safety of two novel malaria vaccines, ChAd63 PvDBP, with or without MVA PvDBP. Heterologous prime-boost with ChAd63-MVA is, to our knowledge, one of the most potent T cell-inducing subunit vaccine regimens which can importantly also induce antibodies. Previous clinical trials using this regimen expressing ME-TRAP, AMA1 & MSP1, have shown that administering ChAd63 as a prime followed 8 weeks later by MVA as a boost is a very immunogenic schedule (32-34). For this reason, and to provide comparability with previous ChAd63-MVA trials, we propose to use a similar administration schedule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner.
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of vaccination.

Agreement to refrain from blood donation during the course of the study.

-Provide written informed consent.

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon.
* History of clinically significant contact dermatitis.
* Any history of anaphylaxis in reaction to vaccination.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg).
* Seropositive for hepatitis C virus (antibodies to HCV) with positive PCR for hepatitis C at screening.
* History of clinical malaria (any species).
* Travel to a malaria endemic region during the study period or within the previous six months.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The safety in healthy volunteers of two new candidate malaria vaccines, ChAd63 PvDBP administered alone, and with MVA PvDBP, in a prime-boost regime. | Up to 20 weeks post first vaccination
  To assess the safety of ChAd63 PvDBP when administered alone and in heterologous prime-boost with MVA PvDBP. Safety will be assessed by the frequency, incidence and nature of adverse events and serious adverse events arising during the study as well as abnormalities in Hematology and Biochemistry lab tests.

SECONDARY OUTCOMES:
The humoral and cellular immunogenicity of ChAd63 PvDBP, when administered to healthy volunteers alone and with MVA PvDBP. | U to 20 weeks post first vaccination.
  PvDBP_RII-specific immunogenicity will be assessed by a variety of immunological assays. These may include ex vivo ELISpot assays for interferon gamma and flow cytometry assays, as well as antibody ELISAs. Other exploratory immunological assays including cytokine analysis, antibody assays, anti-adenovirus antibodies, DNA analysis of genetic polymorphisms potentially relevant to vaccine immunogenicity and gene expression studies amongst others may be performed at the discretion of the investigators.
  Other exploratory immunology may be carried out in collaboration with other specialist labs, including labs outside of Europe. This would involve transfer of serum/plasma, but samples will be anonymised. Volunteers will be consented beforehand.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V S Hill, MD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Payne RO, Silk SE, Elias SC, Milne KH, Rawlinson TA, Llewellyn D, Shakri AR, Jin J, Labbe GM, Edwards NJ, Poulton ID, Roberts R, Farid R, Jorgensen T, Alanine DG, de Cassan SC, Higgins MK, Otto TD, McCarthy JS, de Jongh WA, Nicosia A, Moyle S, Hill AV, Berrie E, Chitnis CE, Lawrie AM, Draper SJ. Human vaccination against Plasmodium vivax Duffy-binding protein induces strain-transcending antibodies. JCI Insight. 2017 Jun 15;2(12):e93683. doi: 10.1172/jci.insight.93683. eCollection 2017 Jun 15. PMID 28614791